CLINICAL TRIAL: NCT00720850
Title: Lenalidomide Maintenance Therapy in Patients With MDS or AML With Cytogenetic Abnormalities Involving Monosomy 5 or del5q After Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Lenalidomide Maintenance Therapy in Patients With Myelodysplastic Syndromes (MDS) or Acute Myelogenous Leukemia (AML)
Acronym: LENAMAINT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment, scientific rationale not applicable anymore to all patients and possible induction of GvHD by the study drug
Sponsor: Technische Universität Dresden (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-LENAMA-022
Record Dates: First submitted 2008-07-17; First posted 2008-07-23 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Myelodysplastic Syndromes; Acute Myelogenous Leukemia
Keywords: MDS; AML; Lenalidomide; monosomy 5; monosomy del5q
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lenalidomide (Experimental): lenalidomide therapy p.o. 10 mg/d for 21 days every 4 weeks for 1 year (12 cycles) after HSCT
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — p.o. 10 mg/d for 21 days every 4 weeks for 1 year (12 cycles) after HSCT
  Other Names: Revlimid

SUMMARY:
The hypothesis of this study is that lenalidomide can be an effective drug in preventing relapse of MDS and AML patients with chromosomal abnormalities involving monosomy 5 or del5q after allogeneic HSCT. Due to its immunomodulatory action it might also be able to enhance a T - or NK cell mediated graft versus leukemia (GVL) effects. Nevertheless, one has to keep in mind a possible, yet unknown influence on modulation of clinical GVHD.

DETAILED DESCRIPTION:
Cytogenetics are main predictors of outcome in patients with MDS and AML. In fact, a monosomy 5 (-5) or del5q (excluding typical 5q-syndrome) are mostly poor prognostic markers also because being frequently part of a complex karyotype. Together, these patients often do not respond to conventional chemotherapy and can only be cured by allogeneic HSCT. Nevertheless, even after transplantation the relapse rate is considerably high and in the majority of patient's relapses occur within the first year after HSCT.

Lenalidomide has been successfully used in MDS patients with del5q, irrespective of additional cytogenetic abnormalities. Furthermore, in vitro studies have demonstrated also impressive anti-proliferative effects of the compound in cell lines harbouring a monosomy 5. Therefore, it seems to be a promising compound in preventing relapse of high-risk MDS or AML patients with chromosomal abnormalities involving del5q or -5 after allogeneic HSCT. Due to its immunomodulatory action it might also be able to enhance T - or NK cell mediated graft versus leukemia effects. Nevertheless, it is unknown whether lenalidomide could modulate or enhance clinical graft versus host disease.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age >=18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* AML (>/= 20% blasts) including secondary (s)AML (after radio-chemotherapy) with karyotype abnormalities involving monosomy 5 or del5q or MDS and sMDS RAEB-1 and RAEB-2 with karyotype abnormalities involving monosomy 5 or del5q or MDS and sMDS type RA(+/-RS) or RCMD(+/-RS) only with complex karyotype abnormalities involving monosomy 5 or del5q
* in complete hematological remission documented by bone marrow aspiration within 8-12 weeks after allogeneic HSCT
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
* ECOG performance status of </= 2 at study entry.
* Laboratory test results within these ranges:

  * Absolute neutrophil count >= 1.0 x 10 9/L
  * Platelet count >= 100 x 10 9/L
  * Serum creatinine <= 2.0 mg/dL
  * Total bilirubin <= 1.5 mg/dL
  * AST (SGOT) and ALT (SGPT) <= 5 x ULN
* Females of childbearing potential (FCBP)† must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed.
* Disease free of prior malignancies for >= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* Able to take aspirin (ASA) 100mg daily as prophylactic anticoagulation in case of concomitant steroid treatment (patients intolerant to ASA may use low molecular weight heparin).

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* active uncontrolled acute GVHD overall grade 3-4
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* History of arterial or venous embolism or stroke
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy to treat MDS or AML within 28 days of baseline (patients within a clinical trial evaluating new conditioning regimens are allowed to participate in the LENAMAINT study)
* Known hypersensitivity to thalidomide or lenalidomide.
* history of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Known positive for HIV or infectious hepatitis, type A, B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of relapse rate | 1 year post transplantation

SECONDARY OUTCOMES:
Overall survival, Incidence and severity of acute and chronic GVHD, Safety | 1 year post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, PD Dr. med., Study Chair — Dresden University of Technology, Medizinische Klinik und Poliklinik 1
Locations (7):
- Germany (7):
  - Dresden University of Technology, Medizinische Klinik und Poliklinik 1, Dresden, Saxony
  - Universitätsklinikum Düsseldorf, Medizinische Klinik und Poliklinik, Klinik für Hämatologie, Onkologie und klinische Immunologie, Düsseldorf
  - Universitätsklinikum Essen, Klinik für Knochenmarktransplantation, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Onkologisches Zentrum, Hamburg
  - Medizinische Hochschule Hannover, Zentrum Innere Medizin, Hämatologie, Hanover
  - Universitätsklinikum Ulm, Klinik für Innere Medizin III, Ulm
  - Universitätsklinikum Würzburg, Medizinische Klinik und Poliklinik II, Würzburg